CLINICAL TRIAL: NCT07097155
Title: Effect of Daily Avocado Consumption on Cellular Aging in Female Breast Cancer Survivors: The ACCA Study
Brief Title: Avocado Consumption and Cellular Aging in Breast Cancer Survivors
Acronym: ACCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Investigacio Sanitaria Pere Virgili (Other)
Responsible Party: Principal Investigator, Nerea Becerra Tomás, Principal Investigator, Institut Investigacio Sanitaria Pere Virgili
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI24/00556
Record Dates: First submitted 2025-07-15; First posted 2025-07-31 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Telomere Length; Breast Cancer Females
Keywords: Avocado consumption; Telomere length; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily Avocado Consumption (Experimental): Participants assigned to the intervention group will be advised to follow their usual diet and to consume one avocado per day for the next four months. To ensure and facilitate compliance with the intervention, we will provide a leaflet with some recipes for incorporating avocados into their regular diet.
  Avocados will be provided for free. Participants will pick up avocados every two weeks from the study site.
  Interventions: Other: Daily Avocado Consumption
- Control - Usual Diet (No Intervention): Participants allocated to the control group will be advised to follow their usual diet. Avocado consumption will not be encouraged.

INTERVENTIONS:
Other: Daily Avocado Consumption — Participants follow their usual diet and consume one avocado per day for 4 months
  Arms: Daily Avocado Consumption

SUMMARY:
Women with breast cancer are at increased risk of comorbidities and premature mortality, potentially due to accelerated biological aging. Telomere attrition has been proposed as a biomarker of this process, which could be mitigated through interventions targeting behavioral factors such as diet. In recent years, avocado has drawn attention in nutritional research due to its unique nutritional profile.

Main objective: To evaluate the effect of consuming one avocado per day on biological aging-measured by telomere length-in breast cancer survivors, compared to a habitual diet (less than two avocados per week). Secondary objectives include changes in telomerase activity and biomarkers of inflammation and oxidative stress. Additional objectives include classical cardiovascular disease markers (glucose metabolism, lipid profile, blood pressure); anthropometric measurements; quality of life and fatigue; and diet quality.

Methodology: A randomized controlled parallel-group trial involving 120 breast cancer survivors. Participants will be randomly assigned to either the intervention group (one avocado per day) or the control group (habitual diet with fewer than two avocados per week) and followed for 4 months. At baseline and the end of the intervention, a general questionnaire will be administered; blood and urine samples will be collected; anthropometric and blood pressure measurements will be taken; and diet, physical activity, quality of life, and fatigue will be assessed. Mean changes from baseline to the end of the intervention in the primary outcome (telomere length) and secondary outcomes (inflammation, oxidative stress, classical cardiovascular disease markers, anthropometric measures, quality of life, and diet) will be compared between the intervention and control groups using linear regression models.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with primary breast cancer in stages I, II or III;
* 40-65 years old at screening;
* Cancer treatment (radiotherapy and chemotherapy) completed ≥ 6 months but not more than 5 years at the time of recruitment;
* Currently consuming less than 2 avocados per week;
* Signed the informed consent letter.

Exclusion Criteria:

* Metastasis;
* Ductal carcinoma or lobular carcinoma in situ;
* Breast cancer recurrence;
* Cancer diagnosis other than breast cancer or non-melanoma skin cancer;
* Body mass index ≥40kg/m2;
* Currently pregnant or breastfeeding, or planning pregnancy in the following 6 months;
* Allergy to latex;
* Unwilling to consume avocado;
* Immunodeficiency or HIV-positive status;
* Alcohol abuse (>50g/day);
* Use of plant sterols, mineral supplements, use of fibre supplements, fish oil, or antioxidants;
* Currently participating in any other randomized controlled trial;
* Difficulty or impossibility of an adequate follow-up;
* Inability or unwillingness to give written informed consent or to communicate with study personnel, or illiteracy;
* Patients with an acute infection or inflammation (e.g., pneumonia) will be allowed to participate in the study 3 months after recovery.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in leukocyte telomere length | Participants will be followed for 4 months. Measurements will be done before and after 4 months.
  Telomere length (TL) analysis will be performed employing the traditional real-time PCR(1) method (Cawthon 2009) by the QuantiTect Syber Green PCR kit (Qiagen). This approach employs the 36B4R single-copy gene as a reference for each sample. The measurements will be performed on a monochrome multiplex real-time quantitative PCR in a BioradCFX96 thermocycler on samples collected before and after the intervention. The data obtained by PCR will be expressed as the ratio of telomere/reference gene (T / S) as the ratio between the number of copies of the telomeric repeat (T) and a single copy gene (36B4F) (S)

SECONDARY OUTCOMES:
Change from baseline in telomerase activity | Participants will be followed for 4 months. Measurements will be done before and after 4 months.
  Telomerase activity will be assessed in white blood cells (PBMCs) using the TeloTAGGG Telomerase PCR ELISAPLUS method, a photometric enzyme immunoassay for quantitative determination of telomerase activity, utilizing the Telomeric Repeat Amplification Protocol (TRAP) (Sigma Aldrich).
Change from baseline in inflammatory markers | Participants will be followed for 4 months. Measurements will be done before and after 4 months.
  Blood samples will be collected in the morning after 8-12h fast. Inflammatory markers (C-reactive protein, IL-1β, IL-6, TNFα, IL-8, IL-10) will be measured by commercial ELISA.
Change from baseline in oxidative markers | Participants will be followed for 4 months. Measurements will be done before and after 4 months.
  Blood samples will be collected in the morning after an 8-12h fast. Oxidized LDL will be measured in plasma.
  Spot urine will be collected, and 8-iso-prostaglandin F2α (8-isoprostanes) will be measured.

OTHER OUTCOMES:
Change from baseline in fasting glucose | Participants will be followed for 4 months. Measurements will be done before and after 4 months.
  Fasting glucose in mg/dL will be measured by standardized methods
Change from baseline in glycated hemoglobin | Participants will be followed for 4 months. Measurements will be done before and after 4 months
  glycated hemoglobin (HbA1c) in % will be measured by standardized methods
Change from baseline in insulin resistance (HOMA-IR) | Participants will be followed for 4 months. Measurements will be done before and after 4 months
  Insulin resistance will be determined by HOMA-IR using plasma glucose and insulin.
Changes from baseline in lipid profile | Participants will be followed for 4 months. Measurements will be done before and after 4 months.
  HDL-cholesterol in mg/dL, LDL-cholesterol in mg/dL, triglycerides in mg/dL, and total cholesterol in mg/dL will be measured
Change from baseline in blood pressure | Participants will be followed for 4 months. Measurements will be done before and after 4 months.
  Systolic and diastolic blood pressure will be measured using an automated device, after 5minutes of resting, in triplicate with a 1-minute interval between each measurement. The first measurement will be discarded, and the average of the two other measurements will be used for analysis.
Change from baseline in body weight | Participants will be followed for 4 months. Measurements will be done before and after 4 months.
  Body weight in kg will be measured, with the participants wearing light clothing and no shoes, using a high-quality electronic scale
Change from baseline in waist circumference | Participants will be followed for 4 months. Measurements will be done before and after 4 months.
  Waist circumference in cm will be measured at the mid-point between the lowest rib and the iliac crest using an anthropometric tape
Change from baseline in BMI | Participants will be followed for 4 months. Measurements will be done before and after 4 months.
  Weight and height will be combined to report BMI in kg/m^2
Change from baseline in body composition | Participants will be followed for 4 months. Measurements will be done before and after 4 months.
  Body composition will be assessed through TANITA
Change from baseline in the Functional Assessment of Cancer Therapy - Breast questionnaire | Participants will be followed for 4 months. Measurements will be done before and after 4 months.
  Quality of life will be assessed through the Functional Assessment of Cancer Therapy - Breast (FACT-B) questionnaire. It is a 37-item instrument designed to measure 5 domains (physical, social, emotional, functional well-being, and breast-cancer subscale) of health-related quality of life in patients with breast cancer.
  Subscale scores will be added to derive:
  1. FACT-B Trial Outcome Index (TOI): ranging from 0 to 96.
  2. FACT-G total score: ranging from 0 to 108
  3. FACT-B total score: ranging from 0 to 148
  The higher the score, the better the outcome.
Change from baseline in the Functional Assessment of Chronic Illness Therapy - Fatigue questionnaire | Participants will be followed for 4 months. Measurements will be done before and after 4 months.
  Fatigue will be assessed through the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) questionnaire, a 40-item measure that assesses self-reported fatigue and its impact upon daily activities and function.
  Subscale scores will be added to derive total scores:
  1. FACIT-F Trial Outcome Index (TOI): ranging from 0 to 108
  2. FACT-G total score: ranging from 0 to 108
  3. FACIT-F total score: ranging from 0 to 160
  4. Fatigue subscale: ranging from 0 to 52
  The higher the score, the better the outcome.
Change from baseline in diet quality | Participants will be followed for 4 months. Measurements will be done before and after 4 months.
  Diet will be assessed using a validated semiquantitative food frequency questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Unit for Public Health and Nutritional Epidemiology, Faculty of Medicine and Health Sciences, Universitat Rovira i Virgili, Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: Undecided